CLINICAL TRIAL: NCT06984432
Title: A Post-marketing, Prospective, Open-label, Single-group, Multicentre Clinical Investigation to Evaluate the Effectiveness and Safety of a Medical Device Based on Non-cross-linked Hyaluronic Acid in Concentrations of 0.55% ("Electri") and 1.1%, 1.8%, or 2.2% ("XELA REDERM") (Diaco Biofarmaceutici S.r.l., Italy) for Improving the Aesthetic Appearance of Facial Skin.
Brief Title: Evaluation of a Non-cross-linked Hyaluronic Acid Medical Device ("Electri" and "XELA REDERM") for Improving Facial Skin Appearance
Acronym: RegHyal-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Hyalual GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Reg.Hyal-01
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Appearance of Facial Wrinkles; Aesthetic; Hydration; Facial Skin Wrinkles
Keywords: facial skin; appearance; hydration; elasticity; XELA REDERM; Electri

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group: Reder malization with Non-Cross-Linked Hyaluronic Acid (Electri and XELA REDERM) (Experimental): Participants in this single-group arm received a course of three redermalization procedures with injectable implants based on non-cross-linked hyaluronic acid. The investigational medical devices included Electri (0.55%) and XELA REDERM (1.1%, 1.8%, or 2.2%), administered intradermally every 14±1 days as part of routine cosmetology practice. The concentration and application area were selected by the investigator based on individual skin conditions. Skin hydration, elasticity, and aesthetic appearance were assessed at baseline and on Days 14, 28, and 42 using instrumental methods and the GAIS scale.
  Interventions: Device: XELA REDERM (non-cross-linked hyaluronic acid 1.1%, 1.8%, or 2.2%); Device: Electri (non-cross-linked hyaluronic acid 0.55%)

INTERVENTIONS:
Device: XELA REDERM (non-cross-linked hyaluronic acid 1.1%, 1.8%, or 2.2%) — Injectable implant containing 1.1%, 1.8%, or 2.2% non-cross-linked hyaluronic acid with succinic acid, sodium succinate, sodium chloride, and water for injection. Intended for redermalization to improve skin quality through biorevitalization.
Device: Electri (non-cross-linked hyaluronic acid 0.55%) — Injectable implant containing 0.55% non-cross-linked hyaluronic acid with succinic acid, sodium succinate, sodium chloride, and water for injection. Intended for redermalization aimed at improving skin hydration, elasticity, and appearance.

SUMMARY:
The goal of this clinical investigation is to learn whether injectable implants based on non-cross-linked hyaluronic acid (Electri and XELA REDERM) improve the aesthetic appearance of facial skin in adult women. It will also learn about the safety of these medical devices.

The main questions it aims to answer are:

Does skin appearance improve after a series of redermalization procedures? How do the procedures affect skin hydration and elasticity? What side effects or medical issues, if any, do participants experience? Researchers did not use a control group. Instead, they evaluated skin improvements in the same participants over time.

Participants:

Received 3 injections of the hyaluronic acid-based device over 6 weeks (1 injection every 14±1 days).

Had their skin condition assessed by doctors and by themselves using a standardized scale.

Underwent tests to measure skin hydration and elasticity. Reported any adverse events or adverse device effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject agreed to participate in the Investigation and signed the Informed Consent Form.
* Age over 18 years.
* The subject is eager to undergo a course of skin redermalization procedures using the medical device(devices) based on non-cross-linked hyaluronic acid in concentrations of 0.55% ("Electri") and 1.1%, 1.8% or 2.2% ("XELA REDERM") (Diaco Biofarmaceutici S. r. l., Italy) in Poland; in concentrations of 1.1%, 1.8% or 2.2% ("XELA REDERM") (Diaco Biofarmaceutici S. r. l., Italy) in Ukraine.
* Female subject confirm that she is not pregnant or lactating during the study.

Exclusion Criteria:

* Infection or inflammation in the implant injection site.
* Pregnancy, lactation.
* Subject's intention to undergo procedures involving chemical peels, laser irradiation, botulinum toxin injection or other similar procedures in the injection site within the next 45 days after inclusion in the post-marketing investigation.
* Subject underwent procedures involving chemical peels, laser irradiation, botulinum toxin injection or other similar procedures in the injection site within 35 days prior to inclusion in the post-marketing investigation.
* Chronic or acute severe or decompensated visceral diseases.
* Known hypersensitivity to hyaluronic acid, its metabolites, or to the excipients of the injectable implant.
* Known hypersensitivity to analgesics.
* Subject took significant doses of vitamin E, NSAIDs or anticoagulants during the last 7 days.
* Refusal or suspected inability of the subject to comply with the requirements of the CIP.
* Subject has difficulty in understanding the language in which the informed consent is written.
* Any other reason that, in the opinion of the investigator, prevents the subject from participating in the post-marketing investigation.
* Subject takes participation in other clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Investigator-assessed improvement in facial skin condition using GAIS scale on Day 42 compared to baseline | Day 42 ±1 after first injection
  The investigator evaluated changes in the aesthetic appearance of facial skin using the Global Aesthetic Improvement Scale (GAIS), a 5-point scale ranging from -1 ("Worse") to 3 ("Very much improved"). The primary endpoint is the mean GAIS score on Day 42 compared to baseline.

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (3):
  - Provita Sp. z o.o., Katowice
  - Ośrodek medyczny OSTEOMED s.c., Krakow
  - Prime Clinic Sp. z o.o., Warsaw
- Institute Hyalual LLC, Kyiv, Ukraine